CLINICAL TRIAL: NCT00326222
Title: Patient Education in NorthTrondelag Hospital Trust - Interventions, Effects and Patient Experience
Brief Title: Patient Education in NorthTrondelag Hospital Trust
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PASOPP1
Record Dates: First submitted 2006-05-15; First posted 2006-05-16 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus
Keywords: Patient Education as a Topic; Self-Management Program; Health promotion; Self Efficacy; Quality of life
MeSH Terms: conditions — Diabetes Mellitus | interventions — Self-Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Lifestyle counseling
  Interventions: Behavioral: Lifestyle counseling
- 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Lifestyle counseling — Self-management group education
  Other Names: Self-management
  Arms: 1

SUMMARY:
The purpose of this randomised open study is to examine the effect of self-management program for diabetes patients.

DETAILED DESCRIPTION:
The primary aim in this study is HbA1c in addition to secondary aims like quality of life and coping.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ICPC-2, code T89 - diabetes dependent on insulin and T90 diabetes not dependent on insulin

Exclusion Criteria:

* Diagnosed with ICPC-2, code T89 - diabetes mellitus juvenile and diabetes I
* Attended self-management program previous 12 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2006-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
HbA1c | Baseline, 6, and 12 mds
PAM - Patient activation measure | Baseline, 6, and 12 mds

SECONDARY OUTCOMES:
SF36 | Baseline, 6, and 12 mds
EQ 5D-VAS scale | Baseline, 6, and 12 mds
Hunt diabetes | Baseline, 6, and 12 mds
WHO-DTSQ | Baseline, 6, and 12 mds
Knowledge of diabetes | Baseline, 6, and 12 mds
HDL-cholesterol | Baseline, 6, and 12 mds
Total cholesterol | Baseline, 6, and 12 mds
Creatinin | Baseline, 6, and 12 mds
Blood pressure | Baseline, 6, and 12 mds
Weight | Baseline, 6, and 12 mds
BMI | Baseline, 6, and 12 mds
Cost/benefit | Baseline, 6, and 12 mds
Triglyceride | Baseline, 6, and 12 mds

CONTACTS AND LOCATIONS:
Overall Officials: Aslak Steinsbekk, PhD, Principal Investigator — Norwegian University of Science and Technology, Trondheim, Norway; Lisbeth O Rygg, Master, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Nord-Trondelag Hospital Trust, Levanger, Nord-Trondelag, Norway

REFERENCES:
- [Result] Rygg LO, Rise MB, Gronning K, Steinsbekk A. Efficacy of ongoing group based diabetes self-management education for patients with type 2 diabetes mellitus. A randomised controlled trial. Patient Educ Couns. 2012 Jan;86(1):98-105. doi: 10.1016/j.pec.2011.04.008. Epub 2011 May 17. PMID 21592715